CLINICAL TRIAL: NCT03742284
Title: Pilot Study to Document Safety and Performance of SoftOx Wound Irrigation Solution in Patients With Split Skin Wounds (Donor Site) Undergoing Skin Transplantation. A Human Model for Acute Trauma Wounds
Brief Title: Safety and Performance of SoftOx Wound Irrigation Solution (SWIS) in Acute Wounds
Acronym: SWIS-01
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: SoftOx Solutions AS (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CIV-18-08-025365
Record Dates: First submitted 2018-11-12; First posted 2018-11-15 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Acute Wounds

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SoftOx Wound Irrigation Solution (Other): SoftOx Wound Irrigation Solution is Medical Device that will be applied to rinse acute wounds.
  Interventions: Device: SoftOx Wound Irrigation Solution

INTERVENTIONS:
Device: SoftOx Wound Irrigation Solution — The SoftOx Wound Irrigation Solution is a Medical device that contains a combination of hypochlorous acid and acetic acid in purified water. SWIS is primary intended for mechanical irrigation of acute wounds whereas hypochlorous acid acts as a ancillary medicinal (drug) substance with potential antimicrobial effects.
  Acute wounds will be rinsed according to protocol and safety (AEs/ADEs/SAEs/SADEs) is the primary objective.
  Other Names: SWIS

SUMMARY:
This pilot study evaluates safety and performance of the Medical device, SoftOx Wound Irrigation Solution (SWIS), in a model for acute wounds.

DETAILED DESCRIPTION:
This is a pilot study with an open-label, exploratory study design with the aim to document preliminary safety and performance of the SoftOx Wound Irrigation Solution while used as intended by the manufacturer, i.e. as an irrigation solution for mechanical rinsing of breached or compromised skin as a result from acute wounds. This first-in-man study will give valuable information on the feasibility of the treatment with the SoftOx Wound Irrigation Solution to prepare for continuous studies in clinically significant settings prior CE marking. The investigation population will consist of 12 subjects undergoing split skin graft transplantation for treating chronic leg ulcers and that are fulfilling the eligibility criteria for the clinical investigation. The SoftOx Wound Irrigation Solution will be applied on the donor site of the split skin graft which is a representative model of acute wounds in a controlled setting. All subjects will be followed up for 21 days. The duration of the investigation is estimated to 4 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 and older
2. Non-healing, leg ulcers, that are scheduled for an operation with excision of the chronic leg ulcer and split skin transplantation
3. Been informed of the nature, the scope and the relevance of the clinical investigation
4. Voluntarily agreed to participation and has duly signed the Informed Consent Form

Exclusion Criteria:

1. Participating in any other clinical investigation
2. On systemic immunomodulating drugs
3. On systemic steroid treatment up to four (4) weeks prior to study inclusion
4. On strong pain medication (e.g. opioids)
5. Severe neuropathy (or dysesthesia on the donor site)
6. Pregnancy
7. Dementia
8. Allergy to polyurethane foam, hypochlorous acid, acetic acid or any other remedies/material used in the clinical investigation
9. Not able to read or understand Danish
10. Any other conditions that as judged by the investigator may make follow-up or investigation inappropriate
11. That according to the Declaration of Helsinki is deemed unsuitable for study enrolment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2018-11-12 (Actual); Primary Completion 2019-05-31 (Estimated); Study Completion 2019-06-15 (Estimated)

PRIMARY OUTCOMES:
- The incidence and severity of any adverse events associated with the SoftOx Wound Irrigation Solution | Evaluation over 21 days
  Incidence and severity of any adverse events related to the SoftOx Wound Irrigation Solution will be summarized in terms of frequencies (n), percentages (%) and the mode.

CONTACTS AND LOCATIONS:
Overall Officials: Ewa A Burian, MD, Principal Investigator — Bispebjerg Hospital
Locations (1):
- Bispebjerg University Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No